CLINICAL TRIAL: NCT05410964
Title: Non-Linear Imaging of Skin In Vivo: VIO In Vivo Skin Imaging evaluatiON (VISION)
Brief Title: Non-Linear Imaging of Skin In Vivo
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: Enspectra Health (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CR-30062; 2R44CA221591-03 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Skin Cancer; Skin Condition; Skin Diseases; Skin Lesion; Skin Abnormalities
MeSH Terms: conditions — Skin Neoplasms; Skin Diseases; Skin Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm
  Interventions: Device: VIO System

INTERVENTIONS:
Device: VIO System — To investigate the potential for the VIO System to display microscopic skin structure in people of different age, sex, race, and skin health

SUMMARY:
The overall objective of this study is to investigate the potential for the VIO System to display microscopic skin structure in people of different age, sex, race, and skin health.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, ages 2 - 90 years old.
2. Subject, or guardian, if applicable, must be willing to provide written informed consent prior to enrollment and agree to comply with protocol requirements. If applicable, child must be willing to provide written assent prior to enrollment and agree to comply with protocol requirements.
3. Subject or guardian, if applicable, must have sufficient mental capacity to understand the Informed Consent and provide clinically relevant and reliable feedback regarding their experience with the device.
4. Subject and guardian, if applicable, must comply with the protocol requirements.
5. Subject or guardian, if applicable, must agree that anonymized personal data will be made available to Study Sponsor and requisite regional and international regulatory bodies.

Exclusion Criteria:

1. Any general health condition or systemic disease that may represent, in the opinion of the Principal Investigator, a potential increased risk associated with device use
2. Currently infected with a communicable skin infection (e.g., shingles or methicillin-resistant S. aureus), which does not include local and minimally pathogenic or non-pathogenic infections distant from the imaging location(s) (e.g., warts, acne)
3. Any known allergies to any materials used in the preparation of skin and/or device use
4. Has a temporary or permanent electrical implanted medical device

   -

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects, volunteers as well subjects with suspected skin condition recruited from dermatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Enspectra Health, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ward WH, Farma JM, editors. Cutaneous Melanoma: Etiology and Therapy [Internet]. Brisbane (AU): Codon Publications; 2017 Dec 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK481860/ PMID 29461771

RESULTS

PARTICIPANT FLOW:
Groups:
- VIO Imaging: Healthy subjects, volunteers as well subjects with suspected skin condition recruited from dermatology clinics
Period: Overall Study
Arm/Group | VIO Imaging
Started | 122
Completed | 122
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VIO Imaging
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 84
  More than one race | 9
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 122
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a demographic measure of skin pigment and sensitivity to sunlight, as self-reported by participants prior to the study procedure. The measure ranges from Type I (least pigment/most sensitive) to Type VI (most pigment/least sensitive). Refer to PubMed ID: 29461771 for the scale used.
  Participants
    Type I | 6
    Type II | 30
    Type III | 46
    Type IV | 25
    Type V | 5
    Type VI | 1
    Unknown | 9
Skin Health [Count of Participants; unit: Participants]
  Healthy | 90
  Suspected or known skin diseases | 32

OUTCOME MEASURES:

1. Primary Outcome: VIO System Imaging Performance
Description: Quantify imaging performance in various types of skin, which may include estimated in vivo resolution and imaging depth. Various types of skin includes skin of different people as well as skin in different locations on the body, and skin with skin disease, including basal cell carcinoma.
  VIO System device design characteristics were iterated during the study to optimize image quality across subjects with various skin types, body locations, and skin disease states. The outcome measure of device imaging performance (acceptable/not acceptable) was assessed through engineering expert review of VIO images. The engineering expert review determined whether images were of consistent quality.
Time Frame: 3 hours
Population: VIO System Imaging Performance assessment was conducted on images taken of all participants
Measure: Number; unit: # participants with acceptable images
Arm/Group | VIO Imaging
Number analyzed (Participants) | 122
# participants with acceptable images | 122

2. Primary Outcome: VIO System Image Quality
Description: Qualitatively evaluate image quality and interpretability by physicians trained in dermatopathology as a function of skin type.
  VIO System device design characteristics were iterated during the study to optimize image quality across subjects with various skin types, body locations, and skin disease states. The outcome measure of device image quality (acceptable/not acceptable) was assessed through clinical expert review of VIO images. The clinical expert review determined whether VIO images could be interpreted by physicians trained in dermatopathology.
Time Frame: 3 hours
Population: VIO System Image Quality assessment was conducted on images taken of all participants
Measure: Number; unit: # participants with acceptable images
Arm/Group | VIO Imaging
Number analyzed (Participants) | 122
# participants with acceptable images | 122

ADVERSE EVENTS:
Time Frame: 1 week
Description: See clinicaltrials.gov definition
Arm/Group | VIO Imaging
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT05410964/Prot_SAP_000.pdf